CLINICAL TRIAL: NCT04121208
Title: A Randomised, Placebo-controlled, Single-blind Study to Characterise the Biomarker Effects of the Colony Stimulating Factor-1 (CSF-1) Receptor Antagonist JNJ-40346527 in Participants With Mild Cognitive Impairment
Brief Title: MIcroglial Colony Stimulating Factor-1 Receptor (CSF1R) in Alzheimer's Disease
Acronym: MICAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Delayed due to COVID19. Study drug expired before could be used.
Sponsor: University of Oxford (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 40346527ALZ1001; 2018-004149-17 (EudraCT Number)
Record Dates: First submitted 2019-07-03; First posted 2019-10-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — JNJ-40346527

STUDY DESIGN:
Intervention Model Description: Phase 1b, randomised, single-blind, placebo-controlled parallel-group trial with JNJ-40346527 in adults with Mild Cognitive Impairment (MCI)
Who Masked: Participant
Masking Description: Single-blind with participants blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug: JNJ-40346527 (Active Comparator): A single initial randomisation site will be set up for Part 1 that will assign participants to JNJ-40346527 300 mg Bis in die - twice a day (BID) or placebo in a 2:1 ratio.
  A second randomisation site will be setup for Part 2 depending on which scenario is adopted.
  Either a "Part 2, Scenario 1" site will assign participants to JNJ-40346527 150 mg BID, JNJ-40346527 50 mg BID or placebo in a 2:2:1 ratio or a "Part 2, Scenario 2" site will assign participants to JNJ-40346527 150-50 mg BID or placebo in a 2:1 ratio.
  Interventions: Drug: JNJ-40346527
- Placebo (Placebo Comparator): Non-active study drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JNJ-40346527 — Active study drug
  Arms: Active drug: JNJ-40346527
Other: Placebo — Non-active study drug
  Arms: Placebo

SUMMARY:
A phase 1 randomised, placebo-controlled, single-blind study to characterise the biomarker effects of the CSF-1 receptor antagonist JNJ-40346527 in participants with mild cognitive impairment. A maximum of 54 participants will be recruited to the two part study. The first part of the study will identify whether it is possible to identify biomarkers that may be used in future studies with JNJ-40346527 and part 2 will investigate a minimal efficacious JNJ-40346527 dose.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a slow, progressive disease that profoundly affects memory and everyday function. There are treatments available that can help manage symptoms, but at present there is no cure, and no treatment that is effective at slowing the progression of AD. AD can begin to cause brain damage decades before symptoms such as memory loss become apparent.

The trial will investigate the effect of the drug JNJ-40346527 on CSF-1R (colony stimulating factor-1 receptor), which is a protein on the outside of cells present in the brain. CSF-1R is responsible for the regulation of various cells, including microglial cells. Recent research suggests that reducing numbers of these microglial cells may be beneficial in slowing the progression of Alzheimer's disease. The Investigators want to see how well JNJ-40346527 is able to block CSF-1R, and in turn suppress these microglial cells. The study is designed to investigate whether or not it is possible to identify changes in levels of proteins which interact with CSF-1R, and changes in the activity or number of affected microglial cells present in the brain. This evidence may provide useful "biomarkers", measures of change in the body, which the Investigators could track to see how the drug is working. These "biomarkers" could then be used in further larger studies to more thoroughly test the benefits of the drug JNJ-40346527. The present study is not designed to test whether or not this drug can slow the progression of Alzheimer's disease.

If biomarkers are identified in the study, further studies will be designed to test whether JNJ-40346527 can slow or prevent the progression of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Any gender over and including 50 years old.
* Willing and able to provide informed consent.
* Clinical Dementia Rating (Scale) (CDR) Global Score = 0.5.
* Self and/or study partner report and impairment on objective cognitive tasks (performance on Hopkin's verbal learning task-revised (HVLT-R) - delay recall and/or free recall > 1 standard deviation (SD) below mean for age/education level).
* Study Partner available, that spends at least 4 hours per week with the participant. The Study Partner must be willing and able to assist with the CDR interview, and will be provided with their own Information Sheet and Informed Consent form.
* Able to read and write in English and with minimum 7 years of formal education.
* Be considered eligible according to the following Tuberculosis (TB) screening criteria:

  1. Have no history of latent or active TB at screening. An exception is made for participants who have a history of latent TB (defined for the purpose of this study as having had a positive result from either the tuberculin skin test or the QuantiFERON-TB® Gold test prior to screening) and documentation of having completed an adequate treatment regimen for latent TB within 1 year prior to the first administration of study agent. Adequate treatment for latent TB is defined according to local country guidelines for immunocompromised patients. If no local guidelines for immunocompromised patients exist, United States (US) guidelines must be followed. It is the responsibility of the Investigator to verify the adequacy of previous anti-TB treatment and provide appropriate documentation.
  2. Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
  3. Have had no recent (within approximately 3 months) close contact with a person with active TB or if there has been such contact, have been evaluated by a physician specialising in TB and found not to have evidence of, or require treatment for latent TB.
* At screening, the results of the following laboratory tests performed at the local laboratory must be within the limits specified below (note: the Investigator may consider the participant eligible if the previously abnormal laboratory test result is within acceptable range on repeat testing. Repeat testing to be done 28 days before dose administration. If results from the laboratory test completed on the same day as the lumbar Puncture are outside the limits specified below, the Investigator may choose to repeat tests and continue the participant in the study, depending on their clinical assessment of any likely outcome/risks).

  1. Haemoglobin ≥8.5 g/dL (International System of Units [SI]: ≥85 g/L)
  2. White Blood Cells (WBC) count ≥3.0 x 103 cells/mm3 (SI:≥ 3.0 x 109 cells/L)
  3. Neutrophils ≥1.5 x 103 cells/mm3 (SI:≥ 1.5 x 109 cells/L)
  4. Lymphocyte count (absolute) ≥450 cells/mm3 (SI: ≥0.45 x 109 cells/L)
  5. Platelets ≥100 x 103 cells/mm3 (SI: ≥100 x 109 cells/L)
  6. Serum alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) levels ≤1.5 x upper limit of normal (ULN)
  7. Total bilirubin levels ≤1.5 x ULN
  8. Serum creatinine ≤1.5 mg/dL
* Be otherwise healthy on the basis of clinical laboratory tests performed at screening. If the results of serum chemistry, haematology, or urinalysis tests not specified in the inclusion criteria above are outside of the normal range, the participant may be included only if the Investigator judges the abnormalities or deviations from normal not to be clinically significant or to be appropriate and reasonable for the population under study.
* A woman, before study entry, must be postmenopausal (amenorrhea for at least 18 months). If a man is heterosexually active with a woman of childbearing potential, he must agree to use a double-barrier method of birth control and not to donate sperm during the study and for 6 months after receiving the last dose of study agent.
* Be willing and able to adhere to all of the procedures, prohibitions and restrictions specified in the protocol.

Exclusion Criteria:

* Research participants who fulfil diagnostic criteria for any type of dementia (e.g. Alzheimer Dementia, Frontotemporal Dementia (FTD), Diffuse Lewy Body Dementia (DLBD), Vascular Dementia (VAD), etc) CDR ≥1.
* Known carriers of a presenilin 1 (PSEN1), presenilin 2 (PSEN2) or Amyloid Precursor Protein (APP) mutation associated with Autosomal Dominant AD or any other neurodegenerative disease.
* Prohibited or restricted concomitant medication as detailed in Section 10.1.7.
* Presence of any neurological, psychiatric or medical conditions associated with a long-term risk of significant cognitive impairment or dementia including but not limited to pre-manifest Huntington's disease, multiple sclerosis, Parkinson's disease, Down syndrome, active alcohol/drug abuse or major psychiatric disorders including current major depressive disorder, schizophrenia, schizoaffective or bipolar disorder. To quantify abuse is to define this as history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-V) criteria within 6 months before screening or positive test result for alcohol and/or drugs of abuse at screening/admission.
* History of latent or active infection of one of the following infectious diseases at screening: Listeria infection, Histoplasma, Coccidioides, Paracoccidioides, Pneumocystis, nontuberculous mycobacteria, Blastomyces, Aspergillus, cytomegalovirus generalised or Herpes zoster infection
* Any cancer or history of cancer in the preceding 5 years (excluding cutaneous basal or squamous cell cancer resolved by excision).
* Any conditions that are clinically significant and may deem the participant's participation in an investigational trial unsafe, e.g., symptomatic cardiovascular disease (including re-vascularisation procedures within the previous year), severe renal or hepatic failure, any clinically relevant abnormalities in blood parameters included in local routine assessments, severe loss of vision, hearing or communicative ability, conditions preventing co-operation or completing the required assessments in the trial, as judged by the Investigator.
* Any contraindications for Lumbar Puncture.
* Any evidence of intracranial pathology which may affect cognition including but not limited to brain tumours (benign or malignant), aneurysm or arteriovenous malformations, territorial stroke (excluding smaller watershed strokes), history of or recovering haemorrhage (parenchymal or subdural), or obstructive hydrocephalus. Research participants with an MRI scan demonstrating markers of small vessel disease (e.g. white matter changes or lacunar infarcts) judged to be clinically insignificant, or microbleeds are allowed.
* Participation in a clinical trial with an Investigational Medicinal Product (IMP) in the last 30 days or 90 days in case of biologics.
* Diminished decision-making capacity that renders the individual not capable of consenting.
* Any other factors in the opinion of the Investigator that could contraindicate the participation of the research participant into this trial.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Placebo-controlled change from baseline in cerebrospinal fluid (CSF) protein marker concentration levels. | Baseline and visit 3 (Days 14)
  Change from baseline in concentration levels of CSF fluid protein markers including but not limited to interleukin (IL)-34 and CSF-1.

SECONDARY OUTCOMES:
Placebo-controlled change from baseline in CSF and blood biomarker concentration levels | Baseline and visit 3 (Days 14)
Placebo-controlled change from baseline in amount of CSF extracellular vesicles and cell population. | Baseline and visit 3 (Days 14)
Measurement of plasma/CSF JNJ-40346527 levels | Baseline and visit 3 (Days 14)
Measurement of cerebrospinal fluid (CSF) protein marker concentration levels following different JNJ-40346527 doses | Baseline and visit 3 (Days 14)
Occurrence of adverse events during the study | Baseline and visit 3 (Days 14). Serious Adverse Events (Day 14 plus 30 days)
  Safety and tolerability will be assessed by monitoring adverse events identified using key safety assessments: physical and neurological examinations, vital sign measurements, clinical laboratory tests and 12-lead ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Raymont, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Cambridgeshire and Peterborough NHS Foundation Trust, Cambridge
  - South London and Maudsley Hospital NHS Foundation Trust, London
  - Oxford Health NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
Study terminated early after 2 participants recruited. No usable data, therefore no data will be shared.